CLINICAL TRIAL: NCT06609993
Title: Thoracic Epidural Analgesia Using Bupivacaine or Ropivacaine With Fentanyl in Patients Undergoing Abdominal Aorctic Repair Under Adequacy of Anaestesia Guidance
Brief Title: AoA Guided Thoracic Epidural Analgesia for Abdominal Aortic Repair
Acronym: AoA-AAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michał Stasiowski (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Sponsor-Investigator, Michał Stasiowski, Principal Investigator, Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Organization: Medical University of Silesia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SilesianMUKOAiIT11
Record Dates: First submitted 2024-08-23; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Aortic Aneurysm; Postoperative Nausea and Vomiting; Postoperative Pain; Haemodynamic Stability
Keywords: Surgical Pleth Index (SPI); General Anaesthesia (GA),; Numerical Pain Rating Scale (NPRS); Adequacy of Anaesthesia (AoA); metamizole; tramadol; thoracic epidural analgesia; bupivacaine; ropivacaine
MeSH Terms: conditions — Aortic Aneurysm; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Operative Blood Salvage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- thoracic epidural analgesia using 0,2% ropicavaine with fentanyl (Experimental): preventive analgesia will be assured using 0,2% ropicavaine (Ropivacaini Hydrochloridum 1%, 10mg/mL, 10 mL, Molteni Farmaceutici, Italy) with fentanyl via thoracic epidural catheter perioperatively
  Interventions: Drug: intravenous rescue opioid analgesia using fentanyl; Drug: intravenous rescue atropine administration; Drug: intravenous rescue urapidil administration; Drug: intravenous rescue ephedrine administration; Biological: concentrate of red blood cells; Biological: red blood cells autotransfusion; Drug: primary treatment of postoperative nausea and vomiting (PONV); Drug: secondary treatment of postoperative nausea and vomiting (PONV); Drug: intraopertative fluid challenge (IFC); Drug: postoperative rescue opioid analgesia using morphine
- thoracic epidural analgesia using 0,2% bupicavaine with fentanyl (Experimental): preventive analgesia will be assured using 0,2% bupicavaine (Bupivacainum Hydrochloricum WZF 0.5%, 5 mg/mL, 10 mL, Polfa Warszawa S.A, Warsaw, Poland) with fentanyl via thoracic epidural catheter perioperatively
  Interventions: Drug: intravenous rescue opioid analgesia using fentanyl; Drug: intravenous rescue atropine administration; Drug: intravenous rescue urapidil administration; Drug: intravenous rescue ephedrine administration; Biological: concentrate of red blood cells; Biological: red blood cells autotransfusion; Drug: primary treatment of postoperative nausea and vomiting (PONV); Drug: secondary treatment of postoperative nausea and vomiting (PONV); Drug: intraopertative fluid challenge (IFC); Drug: postoperative rescue opioid analgesia using morphine
- intravenous analgesia using metamizole with tramadol (Experimental): preventive analgesia will be assured using intravenous infusion using metamizole 5 gram / 24 hours ((Pyralgin 0.5g/ml, 2 ml solution; Polpharma, Poland) with tramadol 400 mg/24h (50 mg/ml, 100 mg/2 ml solution; Polpharma, Poland) perioperatively
  Interventions: Drug: intravenous rescue opioid analgesia using fentanyl; Drug: intravenous rescue atropine administration; Drug: intravenous rescue urapidil administration; Drug: intravenous rescue ephedrine administration; Biological: concentrate of red blood cells; Biological: red blood cells autotransfusion; Drug: primary treatment of postoperative nausea and vomiting (PONV); Drug: secondary treatment of postoperative nausea and vomiting (PONV); Drug: intraopertative fluid challenge (IFC); Drug: postoperative rescue opioid analgesia using morphine

INTERVENTIONS:
Drug: intravenous rescue opioid analgesia using fentanyl — intraoperative rescue opioid analgesia using 1mcg/kg of fentanyl (Fentanyl WZF, POlfa Warsawa, Poland) )/ body weight when SPI value > 15 baseline
  Other Names: IROA-F
Drug: intravenous rescue atropine administration — atropine (Atropinum Sulfuricum WZF, POlfa Warsawa, Poland) in a dose of 0,5mg/kg of will be administered intravenously when heart rate < 50
  Other Names: IRAA
Drug: intravenous rescue urapidil administration — urapidil (Ebrantil 25, Takeda PHARMA, Japan) in a dose of 10 mg will be administered intravenously when DAP > 110 mmHg or SAP > 200 mmHg
  Other Names: IRUA
Drug: intravenous rescue ephedrine administration — ephedrine (Ephedrinum Sulfuricum WZF, POlfa Warsawa, Poland) in a dose of 10 mg will be administered intravenously when DAP < 50 mmHg or MAP < 65 mmHg
  Other Names: IREA
Biological: concentrate of red blood cells — concentrate of red blood cells will be transfused when concentration of haemoglobin < 10g%
  Other Names: RBC
Biological: red blood cells autotransfusion — red blood cells from the operation site will be retransfused using cell saver
  Other Names: cell saver
Drug: primary treatment of postoperative nausea and vomiting (PONV) — dexamethasone ((Dexaven 4mg/ml, Jelfa, Poland) in a dose of 4 mg will be administered intravenously when incidence of PONV is observed
  Other Names: primary treatment of PONV
Drug: secondary treatment of postoperative nausea and vomiting (PONV) — Ondansetron (Ondansetron Accord 2mg/ml, 2 ml solution, Accord Healthcare Limited, Great Britain) in a dose of 4 mg will be administered intravenously when incidence of persistent PONV is observed despite the dexamethasone in a dose of 4 mg will be administration intravenously
  Other Names: treatment of persistent PONV
Drug: intraopertative fluid challenge (IFC) — 3 mililitre of synthetic colloid will be transfused intravenously per each sudden blood loss of 1 mililitre
  Other Names: IFC
Drug: postoperative rescue opioid analgesia using morphine — postoperative rescue opioid analgesia will be administered intravenously using 2 miligrams of morphine ((Morfini Sulfas WZF, 20mg/ml, solutio pro iniectione, Polfa Warszawa, Poland)every 10 minutes until postoperative pain perception using NPRS scale will decrease below 4 (NPRS; 0 meant no pain and 10 meant the worst pain imaginable)
  Other Names: PROA-M

SUMMARY:
The aim of this randomized trial is to assess the efficacy of analgesia using either thoracic epidural or intravenous infusions for open lumbar infrarenal aortic aneurys repair and compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) for monitoring pain perception postoperatively.

Patients received either preemptive thoracic epidural analgesia using either 0,2% ropivacaine with fentanyl or 0,2% bupivacaine with fenthanyl or preemptive intravenous infusion using metamizole and tramadol.

DETAILED DESCRIPTION:
Open major abdominal surgery is one of the most risky surgical procedures performed under general anaesthesia (GA) for inappropriate postoperative pain perception (IPPP), whereas thoracic epidural analgesia (TEA) still constitutes the golden standard of analgesic regimen in the upper abdomen because its was proven to provide improved postoperative analgesia, reduce the incidence of chronic postoperative pain, as compared with parenteral opioids. Therefore, it should always be considered as a routine adjunct to GA for elective open lumbar infrarenal aortic repair (OLIAAR). Monitors of analgesia that measure nociception / antinociception balance - intensity of nociception (painful stimulation) and efficacy of anti-nociception (pain relief) - are increasingly gaining popularity. The Adequacy o Anesthesia (AoA) concept is based on monitoring the depth of GA detected from a forehead sensor using an entropy electroencephalogram (Response Entropy, RE; State Entropy, SE) and the surgical pleth index (SPI) derived from a finger photoplethysmography signal, both of which do not require complex preoperative preparations Observance of the SE value within the range of 40-60 as a result of proper administration of the hypnotic GA component, reflecting the proper suppression of the limbic system, alongside observance of the increase in the SPI value on the monitor (0-no painful stimulation, 100-maximum painful stimulation) after a painful stimulus and returning to the baseline level after the intravenous rescue opioid analgesia (IROA) bolus (anti-nociception), makes the monitoring with AoA guidance easy SPI has been successfully used to monitor analgesia intra- and postoperatively and less postoperative pain have already been reported, when SPI monitoring was employed. Considering all the above, the investigators designed a randomised controlled study to assess the effect of TEA using a combination of either 0,2 % ropivacaine (RPV) and fentanyl (FNT) or 0,2% bupivacaine (BPV) and FNT on intra- and postoperative demand for opioids, haemodynamic stability as compared to intravenous preventive analgesia using metamizole/tramadol in patients undergoing open lumbar infrarenal aortic aneurysm repair (OLIAAR) under AoA-guided GA

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study
* written consent to undergo general anaesthesia combined with different techniques of pre-emptive intravenous or thoracic epidural analgesia for aortic aneurysm repair

Exclusion Criteria:

* antiplatelet therapy
* allergy to local anaesthetics, metamizole or tramadol
* necessity of administration of vasoactive drugs influencing SPI monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
pain perception intraoperatively | from the skin incision till placement of last suture by the operator, an average of 2 hours
  the investigators will compare the efficacy of preventive analgesia intraoperatively according to used preoperatively either intravenous or thoracic epidural infusions . The investigators will administer a rescue dose of fentanyl intravenously in a dose of 1 mcg per kg of body weight in the case when SPI (surgical pleth index) value increases over delta15 points in SPI scale every 5 minutes until SPI value decreases back to baseline value. Additionally, the investigators will analyse rescue fentanyl consumption in abovementioned groups

SECONDARY OUTCOMES:
pain perception postoperatively | from extubation in the operating theatre until discharge to department of vascular surgery, but not shorter than half an hour
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: intravenous infusion of either metamizol/tramadol or thoracic epidural either 0,2% ropivacaine or bupivacaine with fentanyl. The investigators use NPRS (numeric pain rating score 0: no pain - 10: worst possible pain perception) and compare it with SPI values (0: most efficient antinociception-100; worst possible antinociception ).
PONV (postoperative nausea and vomiting) | 48 hours
  The investigators will compare the presence of PONV (scale 0 - no PONV;1 - presence of PONV) after emergence from GA in studied groups. The investigators will observe patients postoperatively for two days and record any incidence of nausea or vomiting and in the abovementioned case the investigators will administer a standard dose of antiemetic drug.
haemodynamic stability | from the beginning of induction of anaesthesia till discharge to department of vascular surgery, on average several hours
  the investigators will observe and note the values of heart rate (HR > 100: tachycardia; < 45: bradycardia) and blood pressure (MAP: mean arterial pressure < 65 mmHg intraoperative hypotension; DAP diastolic arterial pressure > 110mmHg: malignant hypertension)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laferriere-Langlois P, Morisson L, Jeffries S, Duclos C, Espitalier F, Richebe P. Depth of Anesthesia and Nociception Monitoring: Current State and Vision For 2050. Anesth Analg. 2024 Feb 1;138(2):295-307. doi: 10.1213/ANE.0000000000006860. Epub 2024 Jan 12. PMID 38215709
- [Background] Hung KC, Huang YT, Kuo JR, Hsu CW, Yew M, Chen JY, Lin MC, Chen IW, Sun CK. Elevated Surgical Pleth Index at the End of Surgery Is Associated with Postoperative Moderate-to-Severe Pain: A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2022 Sep 6;12(9):2167. doi: 10.3390/diagnostics12092167. PMID 36140567
- [Background] Won YJ, Oh SK, Lim BG, Kim YS, Lee DY, Lee JH. Effect of surgical pleth index-guided remifentanil administration on perioperative outcomes in elderly patients: a prospective randomized controlled trial. BMC Anesthesiol. 2023 Feb 17;23(1):57. doi: 10.1186/s12871-023-02011-5. PMID 36803564
- [Background] Oh SK, Won YJ, Lim BG. Surgical pleth index monitoring in perioperative pain management: usefulness and limitations. Korean J Anesthesiol. 2024 Feb;77(1):31-45. doi: 10.4097/kja.23158. Epub 2023 Mar 17. PMID 36926752
- [Background] Ledowski T, Burke J, Hruby J. Surgical pleth index: prediction of postoperative pain and influence of arousal. Br J Anaesth. 2016 Sep;117(3):371-4. doi: 10.1093/bja/aew226. PMID 27543532
- [Background] Jain N, Gera A, Sharma B, Sood J, Chugh P. Comparison of Surgical Pleth Index-guided analgesia using fentanyl versus conventional analgesia technique in laparoscopic cholecystectomy. Minerva Anestesiol. 2019 Apr;85(4):358-365. doi: 10.23736/S0375-9393.18.12954-3. Epub 2019 Jan 2. PMID 30605991
- [Background] Gold MS, Rockman CB, Riles TS. Comparison of lumbar and thoracic epidural narcotics for postoperative analgesia in patients undergoing abdominal aortic aneurysm repair. J Cardiothorac Vasc Anesth. 1997 Apr;11(2):137-40. doi: 10.1016/s1053-0770(97)90202-0. PMID 9105981
- [Background] Ball L, Pellerano G, Corsi L, Giudici N, Pellegrino A, Cannata D, Santori G, Palombo D, Pelosi P, Gratarola A. Continuous epidural versus wound infusion plus single morphine bolus as postoperative analgesia in open abdominal aortic aneurysm repair: a randomized non-inferiority trial. Minerva Anestesiol. 2016 Dec;82(12):1296-1305. Epub 2016 Aug 30. PMID 27575452